CLINICAL TRIAL: NCT00461942
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Finding Study to Assess the Neuroprotection Effect of Green Tea Polyphenol in De Novo Parkinson's Disease Patients
Brief Title: Efficacy and Safety of Green Tea Polyphenol in De Novo Parkinson's Disease Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Ministry of Health, China (Other Government); Michael J. Fox Foundation for Parkinson's Research (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2004BA702B02-2
Record Dates: First submitted 2007-04-17; First posted 2007-04-18 (Estimated); Last update posted 2011-08-16 (Estimated); Status verified 2011-08

CONDITIONS: Parkinson's Disease
Keywords: Health Food;; Green Tea;; Neuroprotection
MeSH Terms: conditions — Parkinson Disease | interventions — Tea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Green Tea Polyphenols (EGCG/ECG)

SUMMARY:
The purpose of this study is to determine whether Green Tea Polyphenol, an extraction from Green Tea is effective and safe in the treatment of De Novo Parkinson's disease Patients without taking any antiparkinsonism drug

DETAILED DESCRIPTION:
The primary outcome measurement is UPDRS using a delay start design. Total 480 de novo PD patients divided into three dosage groups of green tea polyphenol and one placebo control group. Patients will be treated for one year.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent
* Age 30 years or older at time of diagnosis of Parkinson's disease
* Diagnosed as having typical PD
* Parkinson's disease duration of no more than 5 years
* No current dopaminergic or other forms of anti-parkinsonism therapy
* Hoehn and Yahr stage < 3

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2006-04; Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Delay of progression of Motor dysfunction

SECONDARY OUTCOMES:
Cognition;
Mood;
Quality of Daily life

CONTACTS AND LOCATIONS:
Overall Officials: Piu Chan, MD, PhD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Beijing Institute of Geriatrics, Xuanwu Hospital, Beijing, China